CLINICAL TRIAL: NCT03398096
Title: Improvement of Cardiac Function in Patients With Ischemic Cardiomyopathy by Extracorporeal Shock Wave Therapy: a Multicenter Clinical Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Ya-Wei Xu, Professor, Shanghai 10th People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CSWT
Record Dates: First submitted 2017-12-14; First posted 2018-01-12 (Actual); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cardiac shock wave therapy (CSWT) group (Experimental): The CWST group were performed with a CSWT equipment (Storz Medical, Switzerland) followed the recommended protocol developed by Tohoku University of Japan with respect to the shockwave output and the number of shots implemented to each spot and the protocol developed by the University of Essen, Germany.
  Interventions: Device: Cardiac shock wave therapy
- Control group (No Intervention): No CWST treatment.

INTERVENTIONS:
Device: Cardiac shock wave therapy — Ultrasound guided cardiac shock wave therapy (CSWT) is a new treatment method offering an alternative to revascularization by stimulating angiogenesis. Subsequent clinical trials showed that CSWT could reduce symptoms of myocardial ischemia and improve cardiac function in patients with severe coronary artery disease.
  Arms: Cardiac shock wave therapy (CSWT) group

SUMMARY:
Cardiac shock wave therapy (CSWT) is a noninvasive new therapeutic option in the treatment of chronic refractory angina pectoris. Many domestic and international researches have revealed that CSWT contributes to revascularization by stimulating angiogenesis. We were aimed to evaluate the safety and efficiency of CSWT in the treatment of refractory angina.

ELIGIBILITY:
Inclusion Criteria:

* Patients were 18 to 80 years old;
* Coronary angiography (CA) or multi-slice CT coronary angiography (CTCA) suggestive of moderate to severe coronary artery stenosis;
* Chest tightness, onset of shortness of breath, and poor exercise tolerance after receiving formal drug treatment (with or without stent or bypass graft);
* Hospitalized more than 2 times within 1 year due to the aforementioned problems;
* CCS angina grading higher than grade II, and New York Heart Association (NYHA) class I-III;
* More than 1 month after acute myocardial infarction (AMI) and 1 month after percutaneous coronary intervention (PCI) surgery.

Exclusion Criteria:

* AMI、PCI or coronary artery bypass graft (CABG) within the 4 weeks prior to the study;
* History of heart transplantation;
* History of metal valve replacement surgery;
* Intra-cardiac thrombus;
* Left Ventricular Ejection Fraction (LVEF) < 30 % and unstable hemodynamics;
* Arrhythmia with a rate < 40 bpm or > 120 bpm;
* Skin ulceration or infection in the treatment area;
* Severe obstructive lung disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-03-30 (Estimated); Primary Completion 2018-06-30 (Estimated); Study Completion 2018-09-30 (Estimated)

PRIMARY OUTCOMES:
Canadian Cardiovascular Society (CCS) grading of angina | 6 months
  questionnaire of Canadian Cardiovascular Society grading of angina concerning exercise tolerance
Seattle angina questions (SAQ) | 6 months
  questionnaire of Seattle angina questions to evaluate the effect of coronary artery disease on patients' life quality
6-min walk test | 6 months
  All participants will receive a 6 minutes' walk test to evaluate their effect of treatment of cardiac shock wave therapy
Nitrate consumption | 6 months
  All participants will receive a questionnaire of the amount of nitrate they need before and after treatment of cardiac shock wave therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Weijing L, Ximin F, Jianying S, Mengyun Z, Xuehua F, Yawei X, Liqiong H. Cardiac Shock Wave Therapy Ameliorates Myocardial Ischemia in Patients With Chronic Refractory Angina Pectoris: A Randomized Trial. Front Cardiovasc Med. 2021 Jul 21;8:664433. doi: 10.3389/fcvm.2021.664433. eCollection 2021. PMID 34368242